CLINICAL TRIAL: NCT02383654
Title: An Exploratory Clinical Trial to Assess Treatment of Amyotrophic Lateral Sclerosis With Brain Transplants of Autologous Adipose-Tissue Derived Stem Cells (ADSCs)
Brief Title: Compassionate Treatment : An Exploratory Clinical Trial to Assess Treatment of Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Shinn-Zong Lin, Superintendent, China Medical University Beigang Hospital, Taiwan, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH103-REC2-072
Record Dates: First submitted 2015-02-08; First posted 2015-03-09 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Autologous Adipose-Tissue Derived Stem Cells (ADSCs)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Compassionate Treatment (Other): ALS patients are received Intravenous and intracerebral implantation of Autologous Adipose-Tissue Derived Stem Cells (ADSCs), Rehabilitation.
  Interventions: Procedure: Autologous Adipose-Tissue Derived Stem Cells

INTERVENTIONS:
Procedure: Autologous Adipose-Tissue Derived Stem Cells — 1. Intravenous and Intracerebral implantation of Autologous Adipose-Tissue Derived Stem Cells
  2. Patient will receive brain implantation of approximately 100 -400million Autologous Adipose-Tissue Derived Stem Cells.
  Patient will receive Intravenous of approximately 100-400 million Autologous Adipose-Tissue Derived Stem Cells twice , before brain implantation, and will receive Intravenous of approximately 100-400 million Autologous Adipose-Tissue Derived Stem Cells twice, after brain implantation .
  Other Names: ADSCs

SUMMARY:
The purpose of the study is to determine the safety and possible effectiveness of Autologous Adipose-Tissue Derived Stem Cells treatment in a Amyotrophic Lateral Sclerosis(ALS) patient.

DETAILED DESCRIPTION:
This pilot clinical trial is design to see the safety and possible efficiency of ADSCs treatment in a ALS patient. one subjects will be treated (n=1). The patient will receive brain transplantation of ADSCs and combines intravenous infusion ADSCs 4 times. Subjects will be assessed by adverse effects and functional outcomes of clinical: PI max , PE max,and Haloscale respiration, ALS functional rating scale (ALS-FRS) are analyzed at 1 month, 3 months, 6 months 9 months and 12 months.

Brain MRI scans will be obtained before and after the treatment. Long term follow-up will be performed at 1, 6 , and 12months for safety reasons. Brain CT for check operation safety before and after brain implantation.

Timing of Study: 12months recruitment period after approvals

ELIGIBILITY:
Compassionate Treatment

The number of participants for a person.

The patients (Guo XX) of 28% of lung function assessment (normal lung function was greater than 80%), the daily life of motor function score was 17 points (normal function score of 40 points).

Ages: 35 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
changes of ALS-FRS score | Baseline-Day 28-Day 44-Day 60-6 months-9months-12months
  using ALS-FRS score to assess patient's function after transplantation.
changes of respiratory function | Baseline-Day 28-Day 44-Day 60-6 mouths-9mouths-12mouths
  check the changes of respiratory functions after intervention .
changes of neurologic function | Baseline-Day 28-Day 44-Day 60-6 mouths-9mouths-12mouths
  check any changes of neurologic functions after intervention .

SECONDARY OUTCOMES:
changes of brain structure | Baseline-Day 60- 6 mounths-12 mounths
  check changes of MRI after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shinn-Zong Lin, M.D.;PhD., Principal Investigator — China Medical University Beigand Hospital, Taiwan
Locations (1):
- China Medical University Beigang Hospital, Beigang, Yunlin, Taiwan